CLINICAL TRIAL: NCT02395510
Title: A 10-Week, Open-Label, Flexible Dose Adaptive Study Evaluating the Efficacy of Vortioxetine in Subjects With Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siyan Clinical Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOR-ITT-0024
Record Dates: First submitted 2015-03-16; First posted 2015-03-23 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flexible, open label dosing (Other): Flexible dosing 5-20mg
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine 5-20mg

SUMMARY:
The primary aim of this study is to evaluate the efficacy of Vortioxetine in an adult population with a diagnosis of PD. PD is generally treated with benzodiazepines which are very effective but have a high risk for addiction, fall, and cognitive impairment. There is still a need for better treatment for PD for longer term use. There are other drugs within the SSRI/SNRI class which have proven to be effective in treating patients with this diagnosis.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy of Vortioxetine (5, 10, or 20mg) over a period of 10 weeks in subjects with PD, with or without Agoraphobia. The efficacy of Vortioxetine will be evaluated using the Mean Change from Baseline in the Panic Disorder Severity Scale (PDSS) score and the reduction in occurrence of panic attacks as measured by item 1 in the PDSS Scale after 10 weeks of treatment with Vortioxetine. This study is an open-label, adaptive study with flexible dose strategies lasting 10 weeks. Approximately 20 male and female subjects over the age of 18aged 18-60 years who currently meet DSM-IV criteria for PD with or without Agoraphobia or who have a PDSS score > 8 at Baseline will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily agrees to participate in the study under their own free will.
2. The subject meets the DSM-V criteria for PD with or without Agoraphobia or has a PDSS score > 8 at the Baseline visit.
3. The subject is between the ages of 18-60 years old inclusive at the time of consent.
4. The subject is capable of understanding and complying with protocol requirements.
5. The subject has signed the Informed Consent Form. No study-related procedures may be performed before the subject has signed the form.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing, or may become pregnant during the course of the study. In addition, all subjects of childbearing potential who are sexually active most use adequate contraception from signing of informed consent and throughout the duration of the study. Male subjects who have been surgically sterilized, are at least one year post-vasectomy, are not required to use contraceptives. Females not of childbearing potential are defined as those who have been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (defined as one year since last regular menses).
2. Subjects who have a past or present primary diagnosis with a psychotic disorder other than PD with or without Agoraphobia.
3. Subjects who have a current uncontrolled co-morbid psychiatric disorder other than PD with or without agoraphobia.
4. Subject who have a history of alcohol abuse or dependence within the 12 months prior to screening, as defined by the DSM-V criteria.
5. Subjects who have a comorbid severe medical diagnosis such as Cancer, adults with chronic heart failure, uncontrolled, long-term type 2 Diabetes, etc.
6. Subjects with a history of liver disease such as cirrhosis of liver, neoplasm of the liver, or active Hepatitis C.
7. Subjects weighing less than 100lbs at the Baseline visit.
8. Subjects with a history of cardiac abnormalities including but not limited to, acute cardiovascular events, serious cardiovascular risk, myocardial infarction (MI), unstable angina (UA), percutaneous coronary intervention, coronary artery bypass graft, stroke, or deep vein thrombosis/pulmonary embolism within 1 year of screening, or have planned cardiovascular surgery or percutaneous coronary angioplasty.
9. Subjects who are reasonably judged by the Investigator based on interview or information collected in the Columbia-Suicide Severity Rating Scale (C-SSRS) at the Baseline visit to present a significant suicide risk, or who are likely to require psychiatric hospitalization during the course of the study.
10. Subjects who are unable to fully understand the potential risks and benefits of the study and unable to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in the Panic Disorder Severity Scale (PDSS) score | 10 weeks

SECONDARY OUTCOMES:
Improvement on the Quality of Life Scale (QLOS) from Baseline | 10 weeks
Information from the Monitoring of Side Effects Scale (MOSES) | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Siyan Clinical Corporation, Santa Rosa, California, United States

REFERENCES:
- [Derived] Shah A, Northcutt J. An open-label, flexible dose adaptive study evaluating the efficacy of vortioxetine in subjects with panic disorder. Ann Gen Psychiatry. 2018 May 11;17:19. doi: 10.1186/s12991-018-0190-6. eCollection 2018. PMID 29760763